CLINICAL TRIAL: NCT00811005
Title: Comparison of Fumaric Acid Ester-PUVA (FAE-PUVA) Versus Acitretin-PUVA (Re-PUVA) in Pustular Palmoplantar Psoriasis,a Prospective, Randomized, Controlled, Single-blinded Study
Brief Title: Fumaric Acid Ester-PUVA Therapy Versus Acitretin -PUVA Therapy in Pustular Palmoplantar Psoriasis
Acronym: FVSA-PUVA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Medical University of Vienna / MUW, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-004519-23
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Pustular Palmoplantar Psoriasis
Keywords: acitretin; fumaric acid ester; pustular palmoplantar psoriasis; PUVA
MeSH Terms: interventions — Methoxsalen; 5-Methoxypsoralen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acitretin-PUVA combination (Active Comparator): Acitretin-PUVA combination:
  Acitretin monotherapy: Patients randomized to the acitretin group will receive acitretin in a dose of 1mg /kg daily two weeks prior to additional PUVA treatment.
  PUVA treatment (see below) will be applied thrice weekly in addition to acitretin until (near) complete clearance or over a maximum period of 12 weeks. (Near) complete clearance is defined by improvement of the clinical baseline score (see below) by ≥90%.
  PUVA treatment:
  Intake of 8-methoxypsoralen in a dose of 0.6 mg/kg 1 hour before UVA irradiation or, in case of 8-methoxypsoralen intolerance, 5-methoxypsoralen in a dose of 1.2 mg/kg 2 hours before UVA irradiation.
  Interventions: Radiation: 8-methoxypsoralen or 5- methoxypsoralen; Radiation: 8-methoxypsoralen or 5methoxypsoralen
- Fumaric acid ester -PUVA combination (Experimental): FAE monotherapy:
  Patients randomized to this group will receive FAE in weekly incremental doses (initial daily dose: 30 mg dimethylfumarate (DMF), highest daily dose: 720 mg DMF) starting two weeks prior to additional PUVA treatment.
  FAE-PUVA combination:
  PUVA treatment will be applied thrice weekly in addition to FAE until (near) complete clearance or over a maximum period of 12 weeks. (Near) complete clearance is defined by improvement of the clinical baseline score (see below) by ≥90%.
  PUVA treatment:
  Intake of 8-methoxypsoralen in a dose of 0.6 mg/kg 1 hour before UVA irradiation or, in case of 8-methoxypsoralen intolerance, 5-methoxypsoralen in a dose of 1.2 mg/kg 2 hours before UVA irradiation.
  Interventions: Radiation: 8-methoxypsoralen or 5- methoxypsoralen; Radiation: 8-methoxypsoralen or 5methoxypsoralen

INTERVENTIONS:
Radiation: 8-methoxypsoralen or 5- methoxypsoralen — Intake of 8-methoxypsoralen in a dose of 0.6 mg/kg 1 hour before UVA irradiation or, in case of 8-methoxypsoralen intolerance, 5-methoxypsoralen in a dose of 1.2 mg/kg 2 hours before UVA irradiation.
  Start of PUVA 2 weeks after initiation of acitretin or FAE treatment. Irradiation will be given three times per week over a maximum period of 12 weeks (36 exposures). PUVA exposure will be limited to the hands and feet.
  Other Names: Oxoralen ( 8-methoxypsoralen); Geralen( 5 methoxypsoralen)
Radiation: 8-methoxypsoralen or 5methoxypsoralen — PUVA treatment:
  Intake of 8-methoxypsoralen in a dose of 0.6 mg/kg 1 hour before UVA irradiation or, in case of 8-methoxypsoralen intolerance, 5-methoxypsoralen in a dose of 1.2 mg/kg 2 hours before UVA irradiation.
  Start of PUVA 2 weeks after initiation of acitretin or FAE treatment. Irradiation will be given three times per week over a maximum period of 12 weeks (36 exposures). PUVA exposure will be limited to the hands and feet.
  Other Names: Oxoralen ( 8-methoxypsoralen); Geralen( 5 methoxypsoralen)

SUMMARY:
The purpose of this prospective, randomized, controlled, single-blinded investigation is to study the efficacy, tolerability and safety of oral photochemotherapy (PUVA) combined with acitretin versus oral PUVA combined with systemic fumaric acid esters (FAE) in patients with pustular palmoplantar psoriasis.

Patients will be randomized and allocated in concealed manner to one of the two treatment arms: acitretin-PUVA or FAE-PUVA.

DETAILED DESCRIPTION:
Acitretin-PUVA treatment schedule:

Acitretin monotherapy: Patients randomized to the acitretin group will receive acitretin in a dose of 1mg /kg daily two weeks prior to additional PUVA treatment.

Acitretin-PUVA combination: PUVA treatment (see below) will be applied thrice weekly in addition to acitretin until (near) complete clearance or over a maximum period of 12 weeks. (Near) complete clearance is defined by improvement of the clinical baseline score (see below) by ≥90%.

Acitretin maintenance therapy: After (near) complete clearance patients will be continued on a maintenance dose of 0.5 mg/kg acitretin over 6 months or until significant relapse. Significant relapse is defined by a worsening of the clinical score to ≥50 % of the baseline score.

Follow-up period: Patients who are still significantly improved (clinical score of <50% of the baseline score) will be followed up until significant relapse or over a maximum period of 12 months.

Besides emollients no additional specific treatments will be allowed during the study.

FAE-PUVA treatment schedule:

FAE monotherapy: Patients randomized to this group will receive FAE in weekly incremental doses (initial daily dose: 30 mg dimethylfumarate (DMF), highest daily dose: 720 mg DMF) starting two weeks prior to additional PUVA treatment.

FAE-PUVA combination: PUVA treatment will be applied thrice weekly in addition to FAE until (near) complete clearance or over a maximum period of 12 weeks. (Near) complete clearance is defined by improvement of the clinical baseline score (see below) by ≥90%.

FAE maintenance therapy: After (near) complete clearance FAE will be reduced weekly by 120 mg DMF to a daily maintenance dose of 360 mg DMF which will be administered for a maximum period of 6 months or until significant relapse. Significant relapse is defined by a worsening of the clinical score to ≥50 % of the baseline score.

Follow-up period: Patients who are still significantly improved (clinical score of <50% of the baseline score) will be followed up until significant relapse or over a maximum period of 12 months.

Besides emollients no additional specific treatments will be allowed during the study.

PUVA treatment:

Intake of 8-methoxypsoralen in a dose of 0.6 mg/kg 1 hour before UVA irradiation or, in case of 8-methoxypsoralen intolerance, 5-methoxypsoralen in a dose of 1.2 mg/kg 2 hours before UVA irradiation.

Start of PUVA 2 weeks after initiation of acitretin or FAE treatment. Irradiation will be given three times per week over a maximum period of 12 weeks (36 exposures). PUVA exposure will be limited to the hands and feet.

Primary outcome measure:

Duration of remission

Secondary outcome measures:

Percentage of patients achieving remission Number of PUVA exposures required for inducing remission Total UVA exposure dose required for inducing remission Frequency and quality of adverse reactions

Assessment of clinical response:

A modified local PASI (psoriasis area and severity index) score adapted for the evaluation of the hands and feet will be performed by a blinded investigator at baseline and the onset of PUVA treatment, in biweekly intervals during the course of PUVA treatment, in monthly intervals after discontinuation of PUVA and in bimonthly intervals during a 1-year follow-up period. The study will be terminated in case of a significant relapse which is defined by a PASI score of ≥50 % of the baseline score.

Monitoring:

Prior to the study the blood chemistry, complete blood cell count including differential, urine analysis, TSH, TPO- and TG autoantibodies, a pregnancy tests (in women of childbearing potential) and an ophthalmological examination will be performed. During the study the complete blood cell count, blood chemistry, urine analysis and pregnancy test (in women of childbearing potential) will be reexamined monthly.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pustular palmoplantar psoriasis
* Patients older than 18 years

Exclusion Criteria:

* Pregnant and lactating women
* Uncontrolled hyperlipidemia
* Patients with severely impaired hepatic function
* Patients with severely impaired renal function
* Immunosuppression.
* Abnormal UVA sensitivity
* Intake of photosensitizing drugs
* Oral antipsoriatic therapy within the last 4 weeks
* Topical antipsoriatic therapy within the last 2 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Duration of remission | 12 month

SECONDARY OUTCOMES:
Secondary outcome measures: Percentage of patients achieving remission Number of PUVA exposures required for inducing remission Total UVA exposure dose required for inducing remission Frequency and quality of adverse reactions | 15.5 month

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Tanew, MD, Principal Investigator — Medical University of Vienna; University Clinic of Dermatology
Locations (1):
- Medical University of Vienna; University Clinic of Dermatology; Division of Special and Environmental Dermatology, Vienna, Vienna, Austria